CLINICAL TRIAL: NCT02432391
Title: Self-Monitoring of Blood Glucose (SMBG) as an Educational Tool and a Negative Feedback Loop to Reinforce Blood Glucose Lowering and Discourage Blood Glucose Elevating Self-Management Behaviors in Adults With T2DM
Brief Title: Lifestyle Modification for Type 2 Diabetes Involving Reduction of After-meal Blood Glucose Elevations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: LifeScan (Industry)
Responsible Party: Principal Investigator, Daniel Cox, PhD, Professor, Department of Psychiatry and NB Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16293
Record Dates: First submitted 2015-04-24; First posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Care (No Intervention): Participants continue their routine medical care for type 2 diabetes
- GEM (Experimental): Participants receive the GEM (Glycemic load, Exercise, and Monitoring blood glucose) lifestyle modification program and continue their routine medical care for type 2 diabetes.
  Interventions: Behavioral: GEM

INTERVENTIONS:
Behavioral: GEM — GEM is an integrated lifestyle modification program that focuses on reducing postprandial blood glucose through replacing high with low glycemic load foods and increasing routine physical activity guided by systematic blood glucose monitoring.
  Arms: GEM

SUMMARY:
The purpose of this study is to determine if a lifestyle modification program (GEM) that focuses on reducing after-meal blood glucose elevations can improve blood glucose control in people with type 2 diabetes. Half of the participants will continue their routine medical care, and half will receive five sessions of GEM in addition to their routine care. The two groups will be assessed using diabetes-relevant medical, behavioral and psychological measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes within the past 5 years
* Age >24 and <80 years
* HbA1c >7.0%
* Approval of primary care physician to participate

Exclusion Criteria:

* Currently using, or used within the last 3 months, medications that directly lower BG (e.g., insulin, sulfonylureas, glinides, or DPP-4 inhibitors).
* Currently using, or used within the last 3 months, thiazides at doses above HCTZ 25 mg or equivalent, or loop diuretics above furosemide 20mg or equivalent.
* Currently pregnant or contemplating pregnancy in the coming year
* Currently using, or used within the last 3 months, medications that impede weight loss (e.g., prednisone)
* Having conditions that preclude increasing physical activity, e.g. severe neuropathy, active cardiovascular disease, emphysema, osteoarthritis, stroke.
* Undergoing cancer treatment
* History of lactic acidosis
* Diagnosed with renal impairment

Ages: 24 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline glycosylated hemoglobin at 6 months | 0 and 6 months
  HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cox, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Cox DJ, Fang K, McCall AL, Conaway MR, Banton TA, Moncrief MA, Diamond AM, Taylor AG. Behavioral Strategies to Lower Postprandial Glucose in Those with Type 2 Diabetes May Also Lower Risk of Coronary Heart Disease. Diabetes Ther. 2019 Feb;10(1):277-281. doi: 10.1007/s13300-018-0554-6. Epub 2018 Dec 18. PMID 30565055